CLINICAL TRIAL: NCT04302896
Title: APT-POCT-01: An Open Label, Pharmacokinetic Study of Plasma/Urine/Salivary Drug Concentrations Over Fourteen Days Following Drug Intake Cessation, In HIV-Uninfected Healthy Volunteers Dosing to Steady-state to Further Development of Point of Care Diagnostic Testing
Brief Title: Development of a Urine-Based Point-of-Care Test for Adherence to Antiretroviral Drugs
Acronym: APTAMER
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Rhonda Brand (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor-Investigator, Rhonda Brand, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY19100009; R01AI122301 (NIH)
Record Dates: First submitted 2020-03-06; First posted 2020-03-10 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-03

CONDITIONS: Medication Adherence; HIV
Keywords: Antiretroviral; Pharmacokinetics; Urine Test; HIV negative
MeSH Terms: conditions — Medication Adherence | interventions — dolutegravir; Emtricitabine; tenofovir alafenamide; emtricitabine tenofovir alafenamide; Tenofovir; Lamivudine

STUDY DESIGN:
Intervention Model Description: randomized, open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- dolutegravir + emtricitabine/tenofovir alafenamide (Experimental): Tivicay® (dolutegravir 50 mg tablet) + Descovy® (emtricitabine 200 mg/tenofovir alafenamide 25 mg combination tablet), one tablet of each taken by mouth once daily for 15 days
  Interventions: Drug: dolutegravir oral tablet 50mg; Drug: emtricitabine/tenofovir alafenamide oral tablet 200mg/25mg
- dolutegravir + tenofovir disoproxil fumarate + lamivudine (Experimental): Tivicay® (dolutegravir 50 mg tablet) + Viread® (tenofovir disoproxil fumarate 300 mg tablet) + lamivudine 300 mg tablet, one tablet of each taken by mouth once daily for 15 days
  Interventions: Drug: dolutegravir oral tablet 50mg; Drug: tenofovir disoproxil fumarate oral tablet 300mg; Drug: lamivudine oral tablet 300mg

INTERVENTIONS:
Drug: dolutegravir oral tablet 50mg — Tivicay® (dolutegravir, DTG), a HIV-1 integrase strand transfer inhibitor (INSTI), is FDA-approved in combination with other antiretroviral agents for the treatment of HIV-1 infection in adults and in pediatric patients weighing at least 30kg. Tivicay® 50mg tablets [GlaxoSmithKline] are yellow, round, film-coated, biconvex tablets debossed with "SV 572" on one side and "50" on the other side. The inactive ingredients in each tablet are D-mannitol, microcrystalline cellulose, povidone K29/32, sodium starch glycolate, and sodium stearyl fumarate. The tablet film-coating contains the inactive ingredients iron oxide yellow macrogol/PEG, polyvinyl alcohol-part hydrolyzed, talc, and titanium dioxide.
  Other Names: Tivicay®, DTG
Drug: emtricitabine/tenofovir alafenamide oral tablet 200mg/25mg — Descovy® (emtricitabine/tenofovir alafenamide, FTC/TAF) is a combination of two HIV nucleoside analog reverse transcriptase inhibitors (NRTIs) FDA-approved in combination with other antiretroviral agents for the treatment of HIV-1 infection in adults and pediatric patients weighing at least 35kg. Descovy® 200 mg/25 mg tablets [Gilead] are blue, rectangular-shaped, and film-coated with "GSI" debossed on one side and "225" on the other side. The inactive ingredients are croscarmellose sodium, magnesium stearate, and microcrystalline cellulose. The tablets are film-coated with a coating material containing indigo carmine aluminum lake, polyethylene glycol, polyvinyl alcohol, talc, and titanium dioxide.
  Other Names: Descovy®, FTC/TAF
  Arms: dolutegravir + emtricitabine/tenofovir alafenamide
Drug: tenofovir disoproxil fumarate oral tablet 300mg — Viread® (tenofovir DF, TDF) is a nucleotide analog HIV-1 reverse transcriptase inhibitor and a hepatitis B reverse transcriptase inhibitor FDA-approved for the treatment of HIV-1 infection in combination with other antiretroviral agents and for the treatment of chronic hepatitis B in adults and pediatric patients 2 years of age and older weighing at least 10kg. Viread® 300mg tablets [Gilead] are almond-shaped, light blue, film-coated tablets containing 300 mg of tenofovir disoproxil fumarate, which is equivalent to 245 mg of tenofovir disoproxil, are debossed with "GILEAD" and "4331" on one side and with "300" on the other side. The inactive ingredients in each tablet are croscarmellose sodium, lactose monohydrate, magnesium stearate, microcrystalline cellulose, and pregelatinized starch. Viread® 300mg tablets are coated with Opadry II Y-30-10671-A, which contains FD&C blue #2 aluminum lake, hypromellose 2910, lactose monohydrate, titanium dioxide, and triacetin.
  Other Names: Viread®, tenofovir DF, TDF
  Arms: dolutegravir + tenofovir disoproxil fumarate + lamivudine
Drug: lamivudine oral tablet 300mg — Lamivudine (Epivir®, 3TC) is a nucleoside analogue reverse transcriptase inhibitor FDA-approved in combination with other antiretroviral agents for the treatment of HIV-1 infection in adults and pediatric patients at least 3 months of age. Lamivudine 300mg tablets [Apotex Inc.] are gray, modified diamond-shaped, film-coated, and engraved with "LMV 300" on one side and APO on the reverse side. Inactive ingredients are black iron oxide, colloidal silicon dioxide, crospovidone, hydroxypropyl cellulose, hydroxypropyl methylcellulose, lactose anhydrous, magnesium stearate, polyethylene glycol, and titanium dioxide.
  Other Names: Epivir®, 3TC
  Arms: dolutegravir + tenofovir disoproxil fumarate + lamivudine

SUMMARY:
This is a single-center, open label study to identify adherence levels of commonly prescribed FDA-approved antiretroviral agents by tracking the decline of drug concentrations in plasma, urine and saliva following abrupt drug cessation in HIV-negative adults. Results from this study may provide support for development of a point of care urine testing device to monitor drug adherence.

DETAILED DESCRIPTION:
Poor adherence to antiretroviral (ARV) therapy and HIV pre-exposure prophylaxis (PrEP) incurs costs for patients, health systems, and society. Non-adherence to ARV precedes viral breakthrough and offers opportunities for health-care professionals to intervene. There is a need for accurate, affordable, rapid, and objective monitoring of adherence to be deployed as a companion diagnostic to ARV therapy. Self-reported questionnaires, physician and nurse adherence consistently over-estimate adherence, and pill counts, and pharmacy returns do not yield sufficient precision for individual patients. Therapeutic drug monitoring (TDM) has the advantage tracking medication intake, but sample storage and processing requirements, turnaround times and relatively high cost preclude their widespread deployment. There is a real clinical need for point-of-care adherence testing, which will have high clinical utility by allowing targeting of adherence support and monitoring, better medication review, and integration with community support.

Since the clinical utility of any point-of-care test (POCT) will be its negative predictive value, this trial has been designed as a 'tail' study to track the decline of drug concentrations in plasma, urine and saliva following abrupt drug cessation. Such a study will require dosing to healthy participants who are dosed to steady-state prior to treatment discontinuation.

Serial measurement of drug concentrations in plasma, saliva and urine will be used to develop population-based models which adequately describe the kinetics of elimination and population variability in drug exposure. These models will be used to simulate population drug exposures from which target cut-offs are derived for development of a POCT device.

Approximately thirty healthy, HIV-uninfected participants will be enrolled and equally assigned to one of two ARV dosing arms using a permuted block design randomization scheme.

ARM 1: dolutegravir 50 mg + emtricitabine 200 mg/tenofovir alafenamide 25 mg once daily for 15 days

ARM 2: dolutegravir 50 mg + tenofovir disoproxil fumarate 300 mg + lamivudine 300 mg once daily for 15 days

To assess ARV pharmacokinetics during dosing and over 14 days following ARV cessation, blood, urine, and saliva samples will be collected at Days 1, 2, 8, 15, 16, 17, 18, 19, 22 and 29.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age at screening, verified per site standard operating procedure (SOP)
2. Not pregnant or breastfeeding
3. Availability to return for all study visits, barring unforeseen circumstances
4. Willing and able to

   * communicate in English
   * provide written informed consent to take part in the study
   * provide adequate locator information, as defined in site SOP
   * follow the assigned dosing protocol and maintain an accurate dosing log
5. Must agree not to participate in other concurrent interventional and/or drug trials
6. Understands and agrees to local sexually transmitted infections (STI) reporting requirements
7. HIV-1 seronegative at screening
8. Must be in general good health in the opinion of the investigator
9. For female participants of reproductive potential: Using an effective method of contraception and intending to continue use of an effective method for the duration of study participation and for 8 weeks after the last dose of study drug. Acceptable methods include:

   * hormonal methods
   * IUD (intrauterine device)
   * sterilization of participant or partner

Exclusion Criteria:

1. Participant reports any of the following at Screening:

   1. Has plans to relocate away from the study site area during the period of study participation
   2. Pregnant, less than 3 months post-partum, or lactating
   3. Intends to become pregnant during the period of study participation
   4. History of adverse reaction to study drugs
   5. History of osteoporosis or osteopenia
   6. PrEP (pre-exposure prophylaxis) or (PEP) post-exposure prophylaxis for HIV exposure within 3 months - prior to screening
   7. Participating in another research study involving drugs or medical devices within 3 months or 5 half-lives (if known) prior to enrollment
   8. History of gastric bypass
   9. History of inflammatory bowel disease
   10. Currently taking or anticipation of taking any medications on list of prohibited medications as specified in section 4.10.
   11. Unwilling or unable to comply with study procedures, medications and visits
   12. Allergies to dyes, excipients and components of drugs
   13. Condomless insertive or receptive anal intercourse with more than one partner in the past six months
   14. Known HIV-positive sexual partner within the last 6 months
   15. History of STI in the last 3 months
2. Has any of the following laboratory abnormalities at Screening:

   Note: Grade is per Version 2.1 of the Division of AIDS (DAIDS) Toxicity Table
   1. Hemoglobin Grade 1 or higher
   2. Platelet count Grade 1 or higher
   3. White blood cell count Grade 2 or higher
   4. Calculated creatinine clearance ≤ 70 mL/minute using the Cockcroft-Gault equation
   5. Grade 2 or higher ALT and/or AST (i.e., ≥ 2.5x the site laboratory upper limit of normal [ULN])
   6. Total bilirubin Grade 3 or higher
   7. Positive for Hepatitis B surface antigen (HBsAg)
   8. Confirmed positive for Hepatitis C antibody (HCV Ab)
3. Has any other condition that, in the opinion of the Principal Investigator or designee, would preclude informed consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving study objectives

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Maximum concentration (Cmax) of dolutegravir, emtricitabine, lamivudine, tenofovir disoproxil fumarate, tenofovir alafenamide, and metabolites | Pre-dose; 24, 168, and 336 after the first dose; then 24, 48, 72, 98, 168, and 336 hours after the final dose
  Cmax of dolutegravir, emtricitabine, lamivudine, tenofovir disoproxil fumarate, tenofovir alafenamide, and metabolites in plasma, whole blood (dried spot), saliva, and urine as measured by liquid chromatography tandem mass spectrometry (LC-MS/MS)
Time to maximum concentration (Tmax) of dolutegravir, emtricitabine, lamivudine, tenofovir disoproxil fumarate, tenofovir alafenamide, and metabolites | Pre-dose; 24, 168, and 336 after the first dose; then 24, 48, 72, 98, 168, and 336 hours after the final dose
  Tmax of dolutegravir, emtricitabine, lamivudine, tenofovir disoproxil fumarate, tenofovir alafenamide, and metabolites in plasma, whole blood (dried spot), saliva, and urine as measured by liquid chromatography tandem mass spectrometry (LC-MS/MS)
Minimum concentration (Cmin) of dolutegravir, emtricitabine, lamivudine, tenofovir disoproxil fumarate, tenofovir alafenamide, and metabolites | Pre-dose; 24, 168, and 336 after the first dose; then 24, 48, 72, 98, 168, and 336 hours after the final dose
  Cmin of dolutegravir, emtricitabine, lamivudine, tenofovir disoproxil fumarate, tenofovir alafenamide, and metabolites in plasma, whole blood (dried spot), saliva, and urine as measured by liquid chromatography tandem mass spectrometry (LC-MS/MS)
Area under the concentration-time curve (AUC) of dolutegravir, emtricitabine, lamivudine, tenofovir disoproxil fumarate, tenofovir alafenamide, and metabolites | Pre-dose; 24, 168, and 336 after the first dose; then 24, 48, 72, 98, 168, and 336 hours after the final dose
  AUC of dolutegravir, emtricitabine, lamivudine, tenofovir disoproxil fumarate, tenofovir alafenamide, and metabolites in plasma, whole blood (dried spot), saliva, and urine as measured by liquid chromatography tandem mass spectrometry (LC-MS/MS)
Half-life (t½) of dolutegravir, emtricitabine, lamivudine, tenofovir disoproxil fumarate, and tenofovir alafenamide | Pre-dose; 24, 168, and 336 after the first dose; then 24, 48, 72, 98, 168, and 336 hours after the final dose
  Estimated t½ of dolutegravir, emtricitabine, lamivudine, tenofovir disoproxil fumarate, and tenofovir alafenamide as measured in plasma, whole blood (dried spot), saliva, and urine

CONTACTS AND LOCATIONS:
Overall Officials: Rhonda Brand, PhD, Study Chair — University of Pittsburgh; Ken Ho, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- HIV/AIDS Clinical Research Unit / University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Else LJ, Dickinson L, Edick S, Zyhowski A, Ho K, Meyn L, Dilly-Penchala S, Thompson B, Shaw V, Khoo S, Brand RM. Tenofovir, emtricitabine, lamivudine and dolutegravir concentrations in plasma and urine following drug intake cessation in a randomized controlled directly observed pharmacokinetic trial to aid point-of-care testing. J Antimicrob Chemother. 2024 Jul 1;79(7):1597-1605. doi: 10.1093/jac/dkae147. PMID 38758205

DOCUMENTS (1):
  • Informed Consent Form (2021-02-16): https://cdn.clinicaltrials.gov/large-docs/96/NCT04302896/ICF_000.pdf